CLINICAL TRIAL: NCT05951959
Title: A Multicentre, Phase II, Open-label Study to Evaluate the Efficacy of Acalabrutinib in Combination With Venetoclax and Rituximab in Participants With Treatment Naïve Mantle Cell Lymphoma (TrAVeRse)
Brief Title: A Study of Acalabrutinib Plus Venetoclax and Rituximab in Participants With Treatment Naïve Mantle Cell Lymphoma
Acronym: TrAVeRse
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D822GC00001; 2023-505205-16-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-06-05; First posted 2023-07-19 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Mantle Cell Lymphoma (MCL)
Keywords: Mantle Cell Lymphoma; Lymphoma; Acalabrutinib; Venetoclax; Rituximab
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — acalabrutinib; venetoclax; Rituximab

STUDY DESIGN:
Intervention Model Description: This is a Phase II, open-label, multicentre, international study assessing the efficacy of acalabrutinib in combination with venetoclax and rituximab in adult participants with treatment naïve MCL. Approximately 100 participants with treatment naïve MCL will be treated. The primary objective is to estimate the efficacy of AVR by assessment of CR rate with MRD negativity in participants with treatment naïve MCL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib + Venetoclax + Rituximab (Experimental): Acalabrutinib + Venetoclax + Rituximab (AVR)
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Acalabrutinib — Investigational Product
  Other Names: Acalabrutinib, CALQUENCE
Drug: Venetoclax — Investigator Product
Drug: Rituximab — Investigator Product

SUMMARY:
TrAVeRse is a multicentre, open-label, Phase II study of AVR in treatment naïve MCL participants. The primary objective will be to assess the rate of MRD-negative CR at end of induction after completing 13 cycles of AVR. Participants achieving an MRD-negative CR at the end of AVR induction will be randomised to continued acalabrutinib or observation. Participants who progress during observation may receive retreatment with acalabrutinib

DETAILED DESCRIPTION:
Most mantle cell lymphoma (MCL) patients require treatment at diagnosis. Currently, despite the availability of a number of chemo-immunotherapy-based frontline treatment options, there is no clear superior regimen or curative option for MCL patients. This study aims to evaluate the efficacy of a chemotherapy-free triplet combination regimen of a Bruton's Tyrosine Kinase-inhibitor (acalabrutinib), a BCL2 inhibitor (venetoclax) and an anti-CD20 monoclonal antibody (rituximab) (AVR), in treatment naïve MCL participants.

The study will also assess the feasibility of response-adapted treatment cessation for participants who achieve minimal residual disease (MRD) negative complete response (CR) after AVR induction and the efficacy of retreatment with acalabrutinib in a subgroup of participants who relapse after stopping all anti-lymphoma therapy.

All participants are planned to receive 13 cycles of AVR induction. Each cycle is 28 days. During the induction phase, acalabrutinib is administered twice a day (bd) orally for a total of 13 cycles starting on Cycle 1, venetoclax is administered once daily orally for a total of 12 cycles starting on Cycle 2, and rituximab is administered intravenously on Day 1 of every cycle, for a total of 12 cycles starting on Cycle 1.

* Participants who complete 13 cycles of AVR induction will be centrally tested for MRD status at completion of Cycle 13 and will continue to receive acalabrutinib bd for one full additional cycle (Cycle 14) while awaiting the results of the centralized MRD assessment and evaluation of disease response.
* Participants whose status is MRD-negative CR at the end-of-Cycle 13 assessments will be randomised in a 1:1 ratio to acalabrutinib or observation starting at Cycle 15. Those randomised to acalabrutinib will continue to receive acalabrutinib until progressive disease (PD), death, or unacceptable toxicity whereas those randomised to observation will not receive any anti-lymphoma treatment while in observation. Among the latter group, participants who relapse while in observation may be retreated with acalabrutinib at the time of relapse.
* Participants whose status is MRD-positive CR, PR, or stable disease at the end-of-Cycle 13 assessments will continue to receive acalabrutinib until PD, death, or unacceptable toxicity. The total duration of the study will be approximately 67 months.

Objectives and Endpoints

Primary:

•To assess the efficacy of AVR by assessment of MRD-negative CR rate at the end of AVR induction, i.e., following completion of Cycle 13

Secondary:

* To assess the efficacy of AVR by assessment of MRD-negative CR rate at any time during the study
* To assess the efficacy of AVR by assessment of overall response rate (ORR), CR rate, duration of response (DoR), time to next treatment (TTNT), progression-free survival (PFS), event-free survival (EFS), and overall survival (OS)
* To assess the efficacy of continued acalabrutinib treatment compared to observation, in participants achieving MRD-negative CR after AVR induction by assessment of post randomisation time to first occurrence of relapse or death, EFS, and TTNT
* To assess the safety and tolerability of AVR with continued acalabrutinib or observation until disease progression

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be ≥ 18 years or the legal age of consent in the jurisdiction in which the study is taking place, whichever is greater, at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Histologically documented MCL based on criteria established by the World Health Organization with documentation of chromosomal translocation t(11;14) (q13;q32) and/or overexpression of cyclin D1 in association with other relevant markers (e.g., CD5, CD19, CD20 or PAX5).
3. Clinical Stage II, III, or IV by Ann Arbor Classification and requiring systemic treatment in the opinion of the treating clinician.
4. At least 1 measurable site of disease per Lugano Classification for NHL (Appendix K). The site of disease must be > 1.5 cm in the long axis regardless of short axis measurement or > 1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions, as assessed by diagnostic quality CT (MRI may be used for participants who are either allergic to CT contrast media or have renal insufficiency that per institutional guidelines restricts the use of CT contrast media).

   OR Participant with leukemic non-nodal MCL presentation with splenomegaly (spleen >13 cm in length cranial to caudal) and Bone Marrow (BM) involvement.
5. Eastern Cooperative Oncology Group PS of 0, 1, or 2 and ECOG PS of 3 if poor PS is due to lymphoma.
6. Confirmed availability of sufficient FFPE tumour samples for central laboratory genomic profiling, including TP53 and clone identification for MRD testing per clonoSEQ® assay. Participants with leukemic non-nodal MCL may be enrolled with available BM tissue. For non-nodal leukaemic MCL participants and when nodal or extranodal tissue is not easily accessible and an invasive biopsy will cause a significant risk to the participant, the participant can be enrolled without a tissue biopsy if MCL BM involvement is confirmed by a BM biopsy and sufficient BM biopsy and aspirate provided for TP53 testing, tumour profiling and clone identification for MRD testing.
7. Adequate organ and bone marrow function.

Sex and Contraceptive/Barrier Requirements 8 Male and/or female Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

1. Male participants:

   - Male participants with a female partner of child-bearing potential should use a condom from enrolment, throughout the study until 90 days following the last dose of venetoclax or rituximab, whichever is longer.
   * For non-pregnant potentially childbearing partners, contraception recommendations should also be considered. A male participant must agree to refrain from sperm donation throughout the study until 90 days following the last dose of venetoclax or rituximab, whichever is longer.
2. Female participants:

   * Women of childbearing potential must have negative serum pregnancy test result prior to the start of study intervention (Cycle 1 Day 1) and agree to abstain from breastfeeding during study participation and at least 12 months after the last drug administration.
   * Female participants of childbearing potential who are sexually active with a nonsterilized male partner must agree to use at least one highly effective form of birth control from enrolment, throughout the study and at least 2 days after the last dose of acalabrutinib, at least 6 months after the last dose of venetoclax, and at least 12 months after the last dose of rituximab, whichever is longer.

Informed Consent 9 Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol. Informed consent may be given either by the participant or their legally authorised representative.

10 Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples for optional genetic research that supports the Genomic Initiative.

Exclusion Criteria:

Medical Conditions

1. Active CNS involvement by lymphoma or leptomeningeal disease
2. Current or previous active malignancies requiring anticancer therapy except:

   - adequately treated basal cell or squamous cell skin cancer

   - in situ cancer

   - history of cancer with no evidence of recurrence for ≥ 2 years before enrolment

   - local radiotherapy with a field that does not overlap with sites of current MCL disease and given at least 3 months prior to the screening PET-CT scan and the participant had recovered from any associated toxicity.

   - anti-hormonal therapies are permitted after discussion with the sponsor's medical monitor
3. Participants for whom the goal of therapy is tumour debulking before ASCT
4. Any severe or life-threatening illness, medical condition (e.g., uncontrolled hypertension, bleeding diathesis), or organ system dysfunction which, in the investigator' opinion, could compromise the participant safety, interfere with the absorption or metabolism of study intervention (acalabrutinib, rituximab, venetoclax) or put the study outcomes at undue risk
5. Clinically significant cardiovascular disease such as uncontrolled or untreated symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification, or QTc > 480 msec at screening. Exception: Participants with controlled, asymptomatic atrial fibrillation during screening may enroll.
6. Any active uncontrolled infection (bacterial, viral, fungal, or other infection including tuberculosis), defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment, which in the investigator's opinion makes it undesirable or pose a safety risk for the participant to participate in the study.
7. HIV infection. As per standard of care, results of HIV serology should be known prior to start of study intervention. In the acute situation, registration may occur without the results of the HIV serology but must be available prior to start of study intervention

   Excluded Participants: Participants with active HIV infection (i.e., with detectable viral load by PCR) are excluded.

   Included Participants: HIV-positive participants receiving anti-retroviral treatment with undetectable viral load by PCR may be enrolled following discussion with the participant's HIV physician and the sponsor medical monitor. Potential interactions between anti-retroviral medications and study interventions should be considered.
8. Serologic status reflecting active hepatitis B or C. As per standard of care, results of hepatitis serology should be known prior to start of study intervention. In the acute situation, enrolment may occur without the results of the hepatitis serology but must be available prior to start of study intervention.

   1. Participants who are HBsAg positive or HBV-DNA PCR positive will not be eligible. Participants who are anti-HBc IgG antibody positive and who are HBsAg negative will need to have a negative PCR result before enrolment. Participants who have protective titres of HBsAb after vaccination will be eligible.
   2. Participants who are hepatitis C antibody positive and are HCV-PCR positive will not be eligible.
9. History or ongoing confirmed progressive multifocal leukoencephalopathy.
10. History of stroke or intracranial haemorrhage within 6 months prior to the first dose of study intervention (Cycle 1 Day 1).
11. Uncontrolled autoimmune haemolytic anaemia or idiopathic thrombocytopenic purpura.
12. Active bleeding from a gastrointestinal ulcer, except incidental finding identified on endoscopy that is attributable to MCL
13. Participants with a known hypersensitivity to acalabrutinib, venetoclax, or rituximab or any of the excipients of the product.
14. Known allergy to uric acid lowering agents (e.g., xanthine oxidase inhibitors or rasburicase)
15. Severe prior reactions to monoclonal antibodies
16. Known glucose-6-phosphate dehydrogenase deficiency
17. Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass or inability to swallow the formulated product (tablets).
18. Currently pregnant (confirmed with positive pregnancy test) or breast feeding

    Prior/Concomitant Therapy
19. Any prior therapies for the treatment of MCL with the exception of involved site radiotherapy given at least 3 months prior to screening PET-CT scan and where the radiotherapy field does not overlap areas of current disease activity.
20. Requiring continued treatment with a strong CYP3A4 inhibitor/inducer or its use within 7 days prior to the first dose (Cycle 1 Day 1) of acalabrutinib or venetoclax 21 Requiring continued anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon). Exceptions are DOACs rivaroxaban, apixaban, edoxaban and dabigatran

22 Requiring ongoing immunosuppressive therapy, including systemic or enteric corticosteroids except:

* Topical or inhaled corticosteroids or low-dose oral steroids (≤ 20 mg of prednisone or equivalent per day) as a therapy for comorbid conditions
* Short courses of glucocorticoids in excess of 20 mg prednisone for no more than 14 days for comorbid conditions.
* Systemic use of corticosteroids as a pre-phase to control MCL manifestations (up to approximately 100 mg prednisolone or equivalent daily) for up to 10 days.

  23 Received major surgery (excluding placement of vascular access or for diagnosis) within 28 days of first dose of study intervention (Cycle 1 Day 1) 24 Receipt of live, attenuated vaccine within 28 days before the first dose of study intervention (Cycle 1 Day 1).

See Section 6.9, for lists of prohibited (Table 15) and restricted (Table 16) concomitant medications.

Prior/Concurrent Clinical Study Experience 25 Concurrent participation in another therapeutic clinical trial or participation in another clinical study with an investigational product or investigational medicinal device within 30 days prior to first dose of study treatment (Cycle 1 Day 1).

Other Exclusions 26 Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

27 Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

28 Previous enrolment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2028-07-07 (Estimated); Study Completion 2028-07-07 (Estimated)

PRIMARY OUTCOMES:
MRD-negative CR rate | At the end of AVR induction, i.e., following completion of Cycle 13 (each cycle is 28 days)
  MRD-negative CR rate is defined as the proportion of participants who achieved MRD-negativity in peripheral blood by NGS at a threshold of 10-5 while in CR per the Lugano Classification for NHL at the end of AVR induction

SECONDARY OUTCOMES:
MRD-negative CR rate | Up to approximately 67 months
  MRD-negative CR rate is defined as the proportion of participants who achieved MRD-negativity in peripheral blood by NGS at a threshold of 10-5 while in CR per the Lugano Classification for NHL at any time during the study.
Overall Response Rate (ORR) | Up to approximately 67 months
  ORR is defined as the proportion of participants with a CR or PR, as determined by the investigator.
Overall Response Rate (ORR) | At the end of AVR induction, i.e., following completion of Cycle 13 (each cycle is 28 days)
  ORR is defined as the proportion of participants with a CR or PR, as determined by the investigator.
Complete Response (CR) rate | Up to approximately 67 months
  CR rate is defined as the proportion of participants with a best response of CR.
Complete Response (CR) rate | At the end of AVR induction, i.e., following completion of Cycle 13 (each cycle is 28 days)
  CR rate is defined as the proportion of participants with a best response of CR.
Duration of Response (DoR) | Up to approximately 67 months
  The DoR is defined as the time from the date of first documented response (CR-PR) until the date of documented progression per the Lugano Classification for NHL or death (by any cause in the absence of disease progression), whichever occurs first.
Time to Next Treatment (TTNT) | Up to approximately 67 months
  TTNT or death is defined as the time from the start of AVR induction until the start of the next anti-lymphoma therapy (including local radiotherapy, unless pre-planned at baseline) or death due to any cause, whichever comes first.
Progression-free Survival (PFS) | Up to approximately 67 months
  PFS is defined as the time from the start of AVR induction until the date of documented objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from therapy or receives another anti-cancer therapy prior to progression.
Event Free Survival (EFS) | Up to approximately 67 months
  EFS is defined as the time from the start of AVR induction to any of the following events: disease progression, or initiation of systemic anti-lymphoma treatment and or unplanned radiation, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 67 months
  OS is defined as the time from the start of AVR induction until death due to any cause.
Post randomization time to first occurrence of relapse or death, EFS and TTNT in continued acalabrutinib arm compared to observation arm. | Yearly from Cycle 15 (each cycle is 28 days) Day 1, until 3 years after randomization
  Time to first occurrence of relapse or death is defined as the time from Cycle 15 Day 1 until date of progression per the Lugano Classification for NHL as assessed by investigator, or death due to any cause, whichever occurs first.
  Event-free survival is defined as the time from Cycle 15 Day 1 until any of the following events: disease progression, or initiation of subsequent systemic anti-lymphoma treatment and/or unplanned radiation, or death due to any cause, whichever occurs first.
  Time to next therapy or death is defined as the time from Cycle 15 Day 1 until the start of the next anti-lymphoma therapy (including local radiotherapy, unless pre-planned at baseline) or death due to any cause, whichever comes first.
Number of participants with any Adverse Events (AE), Serious Adverse Events (SAE), Adverse Event of Special Interest (AESI) and AEs leading to study treatment discontinuation or dose modification. | Up to approximately 67 months
  Adverse events will be graded by the investigator according to the NCI-CTCAE v5.0. Each AE verbatim term will be coded to a system organ class and a preferred term using the MedDRA.

CONTACTS AND LOCATIONS:
Locations (28):
- United States (5):
  - Research Site, Hackensack, New Jersey
  - Research Site, Stony Brook, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
- Australia (4):
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Nedlands
  - Research Site, Sydney
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Poland (3):
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Warsaw
- Research Site, Madrid, Spain
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Gloucester
  - Research Site, London
  - Research Site, Norwich
  - Research Site, Nottingham
  - Research Site, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided